CLINICAL TRIAL: NCT04867252
Title: Effects of Combined Resveratrol and Myo-inositol on Altered Metabolic, Endocrine Parameters and Perceived Stress in Patients With Polycystic Ovarian Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Mohsin Shah, Associate Professor, Khyber Medical University Peshawar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASRB001226/EC/IBMS
Record Dates: First submitted 2021-04-24; First posted 2021-04-30 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: PCOS
Keywords: PCOS, Resveratrol and Myoinositol
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Resveratrol; Inositol; Metformin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Therapy Group (Active Comparator): ARM 1: Resveratrol (1000mg Twice a day) Myoinositol (1000mg Twice a day)
  Interventions: Drug: Resveratrol (1000mg twice a day), Myoinositol 1000mg (Twice a day)
- Standard Therapy Group (Other): ARM 2:Metformin 500mg (Twice a day) Pioglitazone (15mg Twice a day)
  Interventions: Drug: Metformin (500 mg Twice a day), Pioglitazone (15 mg Twice a day)

INTERVENTIONS:
Drug: Resveratrol (1000mg twice a day), Myoinositol 1000mg (Twice a day) — 51 Patients with PCOS receiving Resveratrol and Myoinositol 1000mg and 1000mg BD daily respectively
  Arms: Combination Therapy Group
Drug: Metformin (500 mg Twice a day), Pioglitazone (15 mg Twice a day) — 51 Patients with PCOS receiving Metformin and Pioglitazone 500 mg and 15 mg BD daily respectively
  Other Names: Zolid Plus
  Arms: Standard Therapy Group

SUMMARY:
The investigators aim is to conduct a double blind randomized clinical trial, to study the effects of combined Resveratrol and Myo-Inositol on altered metabolic, endocrine parameters and perceived stress response in patients with Polycystic Ovary Syndrome (PCOS). Women diagnosed with PCOS, using criteria proposed in November 2015, by the American Association of Clinical Endocrinologists (AACE), American College of Endocrinology (ACE), and Androgen Excess and PCOS Society (AES) for PCOS should include two of the following three criteria: chronic an ovulation, hyperandrogenism (clinical/biologic), and polycystic ovaries. The investigators propose that PCOS women may have altered metabolic, endocrine levels and increased perceived stress response and combination therapy may have beneficial influences on these parameters in women diagnosed with PCOS.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) is extremely prevalent and considered to be the most common heterogeneous endocrine disorder in reproductive age women. This affects up to 10-15% of women in reproductive age. PCOS is a multifaceted health issue characterized by chronic anovulation with excess ovarian activity, hyperandrogenism and polycystic ovaries. The most disappointment for women with PCOS is pregnancy loss.

This endocrine disorder has some long term effects including cardiovascular diseases, metabolic and sexual dysfunction, depression and anxiety that effects the overall quality of life. Women with PCOS have a greater risk of developing hyperinsulinemia and insulin resistance and this explains the substantially increased prevalence of glucose intolerance in PCOS. Recent long-term follow up studies of the syndrome have shown that dyslipidemia and hyperlipidemia is a very common metabolic abnormality in these women. The key pathophysiology of PCOS is Insulin resistance, thus dyslipidemia in women may be constant with those found in an insulin resistant state. Low adiponectin levels in PCOS have been largely associated with obesity which is common among these patients. Serum adiponectin levels are associated with PCOS independently and are only explained by IR partly. An independent biomarker, adiponectin can be used for diagnosing PCOS in young and lean women or women with a family history of PCOS.

Resveratrol (3,5,4-trihydroxy-trans-stilbene) belongs to polyphenols stilbene group found in grapes, peanuts, red wine and many medicinal plants. Studies have shown that patients treated with resveratrol have shown improve glucose homeostasis and reverse insulin resistance. Treatment with resveratrol improved the elevated number of atretic and secondary follicles and the decreased number of Graafian follicles in the PCOS group, which indicates the effect of the treatments on the maintenance of folliculogenesis. It has been reported to interact with multiple cell targets, but its major effects are brought about by the activation of SIRT1 (silent information regulator1).The SIRT1 is expressed in oocytes and human granulosa nuclei cells at multiple developmental stages of the follicles. It is also responsible for suppressing inflammation. Moreover, SIRT1 is also involved in protecting the oocytes from age dependent insufficiencies through oxidative stress.

Myo-Inositol is a carbocyclic sugar, belongs to Inositol group and is an important component of structural lipids. Inositol's or its phosphates and the associated lipids are found in different fruits specially cantaloupe and oranges. It is the precursor of inositol triphosphate, acting as an intracellular second messenger and regulating a number of hormones such as thyroid-stimulating hormone, follicle-stimulating hormone (FSH) and insulin. One of the insulin-sensitizing compounds, Myo-Inositol is capable of restoring spontaneous ovarian activity, and consequently fertility, in most patients with PCOS. Inositol's improve the metabolic and endocrine parameters in young, overweight PCOS patients and regulate the monthly cycles. Treatment with inositol's in obese PCOS patients is also effective in reducing BMI. The decrease in BMI is without any lifestyle modification.

PCOS is a systemic condition, an endocrinopathy whose etiology is still not understood, correct treatment regimens of PCOS will not only improve menstrual cycles of the patients but will also improve the metabolic or endocrinological parameters. PCOS sufferers are also known to have increased levels of perceived stress which will be considered in the study. Very little evidence is available on combination therapy for treatment of PCOS patients. In this study our goal will be to come up with a better treatment option to treat the disease effectively.

Study Objectives:

To investigate the effects of combined Resveratrol and Myo-Inositol treatment after 3 months on metabolic, endocrine alterations and perceived stress response in patients with PCOS.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment naive PCOS women having age from 14-45 years with scanty or no menstruation, hirsutism and elevated serum androgen levels, will be diagnosed on the basis of AES (Androgen access society) guidelines 2006 according to which when two of the following criteria are present patient will be said to have the syndrome
2. Hirsutism or hyperandrogenism
3. Oligo or an-ovulation and or polycystic ovaries

Exclusion Criteria:

1. Women with previous history of Cushing syndrome
2. Thyroid disorders
3. Hyperprolactinemia
4. Ovarian tumors
5. Congenital adrenal hyperplasia androgen-producing tumors,
6. History of seizures
7. Patients on warfarin, Coumadin and Sintrom because of drug interaction with acetyl-L-Carnitine,
8. Pregnancy or using contraceptive medications,
9. Patients on hormonal therapy that alters the biochemical or hormonal profile

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance | 3 months
  PCOS associated insulin resistance and hyperinsulinemia through HOMA-IR
Hypoadiponectinemia | 3 months
  PCOS associated Hypoadiponectinemia. Measurement of adiponectin levels through human adiponectin enzyme-linked immunosorbent assay (ELISA ) kit and the values of serum adiponectin reported in microgram/mL.
Ovary volume | 3 months
  Polycystic ovaries volume measurement by abdominopelvic ultrasound
Stress response | 3 months
  Perceived stress response and profile of mood stress by structured questionnaire

SECONDARY OUTCOMES:
Body fat analysis | 3 months
  Body fats measurement through measurement scale
Hirsutism | 3 months
  Hirsutism grading scale, Ferriman Gallwey Score is used to evaluate hirsutism. A score of 1 to 4 is given for nine areas of the bod including upper lip, chin, chest, upper abdomen, lower abdomen, arms, thighs, upper back and lower back. A total score less than 8 is considered normal, a score of 8 to 15 indicates mild hirsutism, and a score greater than 15 indicates moderate or severe hirsutism. A score of 0 indicates absence of terminal hair.
Abnormal menstruation patterns both oligomenorrhea or amenorrhea attributed to chronic anovulation | 3 months
  Oligomenorrhea evaluated by menstrual bleeding that has occurred at intervals of 35 days to 6 months, with < 9 menstrual periods per year and secondary amenorrhea assessed by absence of menstruation for 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mohsin Shah, PhD, Principal Investigator — Department of Physiology, Khyber Medical University, Peshawar Pakistan
Locations (1):
- Gynecology and Obstetric, Hayatabad Medical Complex, Peshawar, Khyber Pukhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rocha AL, Oliveira FR, Azevedo RC, Silva VA, Peres TM, Candido AL, Gomes KB, Reis FM. Recent advances in the understanding and management of polycystic ovary syndrome. F1000Res. 2019 Apr 26;8:F1000 Faculty Rev-565. doi: 10.12688/f1000research.15318.1. eCollection 2019. PMID 31069057
- [Background] Monastra G, Unfer V, Harrath AH, Bizzarri M. Combining treatment with myo-inositol and D-chiro-inositol (40:1) is effective in restoring ovary function and metabolic balance in PCOS patients. Gynecol Endocrinol. 2017 Jan;33(1):1-9. doi: 10.1080/09513590.2016.1247797. Epub 2016 Nov 29. PMID 27898267
- [Background] Sirmans SM, Pate KA. Epidemiology, diagnosis, and management of polycystic ovary syndrome. Clin Epidemiol. 2013 Dec 18;6:1-13. doi: 10.2147/CLEP.S37559. PMID 24379699
- [Background] Carmina E, Lobo RA. Polycystic ovary syndrome (PCOS): arguably the most common endocrinopathy is associated with significant morbidity in women. J Clin Endocrinol Metab. 1999 Jun;84(6):1897-9. doi: 10.1210/jcem.84.6.5803. No abstract available. PMID 10372683
- [Background] Bajuk Studen K, Pfeifer M. Cardiometabolic risk in polycystic ovary syndrome. Endocr Connect. 2018 Jul;7(7):R238-R251. doi: 10.1530/EC-18-0129. Epub 2018 May 29. PMID 29844207
- [Background] Dunaif A. Insulin resistance and the polycystic ovary syndrome: mechanism and implications for pathogenesis. Endocr Rev. 1997 Dec;18(6):774-800. doi: 10.1210/edrv.18.6.0318. PMID 9408743
- [Background] Kim JJ, Choi YM. Dyslipidemia in women with polycystic ovary syndrome. Obstet Gynecol Sci. 2013 May;56(3):137-42. doi: 10.5468/ogs.2013.56.3.137. Epub 2013 May 16. PMID 24327994
- [Background] Mirza SS, Shafique K, Shaikh AR, Khan NA, Anwar Qureshi M. Association between circulating adiponectin levels and polycystic ovarian syndrome. J Ovarian Res. 2014 Feb 7;7:18. doi: 10.1186/1757-2215-7-18. PMID 24502610
- [Background] Salehi B, Mishra AP, Nigam M, Sener B, Kilic M, Sharifi-Rad M, Fokou PVT, Martins N, Sharifi-Rad J. Resveratrol: A Double-Edged Sword in Health Benefits. Biomedicines. 2018 Sep 9;6(3):91. doi: 10.3390/biomedicines6030091. PMID 30205595
- [Derived] Hassan S, Shah M, Malik MO, Ehtesham E, Habib SH, Rauf B. Treatment with combined resveratrol and myoinositol ameliorates endocrine, metabolic alterations and perceived stress response in women with PCOS: a double-blind randomized clinical trial. Endocrine. 2023 Jan;79(1):208-220. doi: 10.1007/s12020-022-03198-2. Epub 2022 Sep 28. PMID 36169918